CLINICAL TRIAL: NCT01355861
Title: Negative Work Exercise as a Novel Treatment for Sarcopenia in Older Men
Brief Title: Resistance Exercise for the Prevention of Age-related Sarcopenia
Acronym: REPAiRS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Project has been withdrawn from funding consideration
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Harris-Love, Michael - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E7508-W
Record Dates: First submitted 2011-03-14; First posted 2011-05-18 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Sarcopenia
Keywords: sarcopenia; aging; rehabilitation; exercise
MeSH Terms: conditions — Sarcopenia; Motor Activity | interventions — Cadaverine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Exercise group 1: Negative work exercise
  Interventions: Behavioral: Negative work exercise
- 2 (Other): Exercise group 2: Negative work exercise (delayed start for single-arm crossover trial)
  Interventions: Behavioral: Negative work exercise

INTERVENTIONS:
Behavioral: Negative work exercise — Submaximal negative work exercise using an isokinetic dynamometer will be performed twice per week for 12 weeks. Exercise volume will be 3 sets of 10 repetitions for the knee and shoulder extensors.
  Other Names: Biodex

SUMMARY:
The purpose of this study is to determine the benefits of negative work progressive resistance exercise (PRE) for the conservative management of sarcopenia in older male Veterans at the DC VAMC. Efficacy will be assessed by examining post-exercise changes in metabolic and inflammatory markers, muscle morphology, strength, and functional status.

DETAILED DESCRIPTION:
The chief aim of this protocol is to determine the efficacy of negative work progressive resistance exercise (PRE) in the management of sarcopenia in older male Veterans at the DC VAMC. This proposed study is a randomized clinical trial using a single-arm, delayed cross-over design with repeated measures. This method is a patient-first approach to clinical research that permits all participants to receive the intervention while allowing the investigators to conduct both within subjects and between subjects comparisons with a modest study enrollment. During the "pre-treatment period" we will recruit, screen, and consent 30 older men with sarcopenia. The participants will be randomized into two groups: active treatment and delayed treatment. The initial "active treatment" and "delayed treatment" periods will last 12 weeks. After 12 weeks, the participants in the delayed treatment group will crossover (without a washout period) and start 12 weeks of intervention. All participants will detrain and be monitored for follow up during their respective 12-week "post treatment" period. Outcome measures include post-exercise changes in metabolic and inflammatory markers, muscle morphology, strength, and functional status.

ELIGIBILITY:
Inclusion Criteria:

Adult, ambulatory males > 60 years old (n=30) will be recruited for this proposed study. Participant inclusion criteria also includes having clinically significant sarcopenia based on the body composition assessment showing an aLM that is < 2 SD below the mean values of a young adult reference group using DEXA scanning.

Exclusion Criteria:

Exclusion criteria include BMI scores > 30 or a Mini-Mental Status exam score of < 22. The second tier of screening will include the following blood tests, obtained between 8-9 AM, following a 12-hour overnight fast: CBC, routine chemistry profile (e.g., glucose, kidney and liver function tests). Veterans with an elevated fasting blood glucose by WHO criteria (FBG >110 mg/dl), triglyceride levels > 200 mg/dL, and/or known DM, or abnormalities of other routine blood tests (i.e., > 2 SD beyond normal) will be excluded from the study. Uncontrolled cardiovascular disease, non-ambulatory status, evidence of a major disease exacerbation over the last six months, and current participation in a supervised exercise program (minimum of three months, twice per week) would also preclude participation in this study.

Ages: 60 Years to 79 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Changes in insulin sensitivity following the exercise intervention as estimated with the QUICKI algorithm (quantitative insulin sensitivity check index) | Change from baseline in QUICKI values at week 6, week 12, and week 24
  Blood tests will be obtained after a 12- hour overnight fast at baseline, weeks 6, week 12 and week 24: glucose and insulin values will be determined before and during a standard (75 g) 2 hour oral glucose tolerance test (to determine insulin sensitivity via QUICKI algorithm.

SECONDARY OUTCOMES:
Peak isokinetic torque | Treatment weeks: 1, 6, and 12; post-treatment weeks: 6 and 12
  Isokinetic knee and shoulder extension torques will be obtained bilaterally using the Biodex System 3
Diagnostic ultrasongraphy | Treatment weeks: 1, 6, and 12; post-treatment weeks: 6 and 12
  Muscle thickness, pennation angle, and area at the flexor digitorum superficialis, lower-trapezius, rectus femoris and tibialis anterior (dominant side only).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Harris-Love, DSc MPT BS, Principal Investigator — VA Medical Center, DC
Locations (1):
- VA Medical Center, DC, Washington D.C., District of Columbia, United States